CLINICAL TRIAL: NCT00600444
Title: Randomized Controlled Trial Comparing Venae Sectio Versus Punction of Vena Subclavia for Insertion of a Totally Implantable Access Port
Brief Title: PORTAS 2, Comparing Venae Sectio Versus Punction of Vena Subclavia for Insertion of a Totally Implantable Access Port
Acronym: PORTAS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. med. M. W. Büchler, Chairman Department of Surgery, University of Heidelberg, Department of General, Visceral and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSC01/08
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-05

CONDITIONS: Cancer
Keywords: permanent venous access; chemotherapy; parenteral nutrition; Patients with a benign and/or malignant diseases which demand a safe and permanent venous access, e.g. for chemotherapy and/or parenteral nutrition; benign diseases; malignant diseases
MeSH Terms: conditions — Neoplasms; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Venae Sectio technique will be used to insert totally implantable access port (TIAP) by a surgeon
  Interventions: Procedure: Venae sectio
- B (Experimental): Punction of Vena Subclavia will be used to insert totally implantable access port (TIAP) by a radiologist.
  Interventions: Procedure: Punction of V. subclavia

INTERVENTIONS:
Procedure: Venae sectio — surgical preparation of the cephalic vene to insert a totally implantable access port.
  Arms: A
Procedure: Punction of V. subclavia — radiological punction of the v. subclavia with Seldinger technique to implant a totally implantable access port
  Arms: B

SUMMARY:
The purpose of this trial is to investigate if the success rate of punction the vena subclavia (99% in retrospective studies) will be 15% higher than the success rate of venae sectio (80% in retro and prospective studies) for implantation of a totally implantable access ports.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years
* Patients scheduled for primary elective implantation of TIAP

Exclusion Criteria:

* Participation in another clinical trial which could interfere with the primary endpoint of this study
* Lack of compliance
* Impaired mental state or language problem
* Patients with known allergy to contrast agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Primary success rate of the randomized intervention | Assessed on the day of surgery (day 0)

SECONDARY OUTCOMES:
Peri-/postoperative complication rate for the randomized intervention | Assessed after 90 day post operation

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Büchler, Prof. Dr., Principal Investigator — University of Heidelberg, Department of General, Visceral and Transplantation Surgery
Locations (1):
- University of Heidelberg, Heidelberg, Baden Würtemberg, Germany

REFERENCES:
- [Derived] Knebel P, Lopez-Benitez R, Fischer L, Radeleff BA, Stampfl U, Bruckner T, Hennes R, Kieser M, Kauczor HU, Buchler MW, Seiler CM. Insertion of totally implantable venous access devices: an expertise-based, randomized, controlled trial (NCT00600444). Ann Surg. 2011 Jun;253(6):1111-7. doi: 10.1097/SLA.0b013e318214ba21. PMID 21412146
- [Derived] Knebel P, Fischer L, Cremonese E, Lopez-Benitez R, Stampfl U, Radeleff B, Kauczor HU, Buchler MW, Seiler CM. Protocol of an expertise based randomized trial comparing surgical Venae Sectio versus radiological puncture of Vena Subclavia for insertion of Totally Implantable Access Port in oncological patients. Trials. 2008 Oct 24;9:60. doi: 10.1186/1745-6215-9-60. PMID 18950491